CLINICAL TRIAL: NCT06739837
Title: Comparison of the Effect of a Non-immersive Virtual Reality Environment and Conventional Treatment in Patients With Tennis Elbow
Brief Title: Comparison of the Effect of a Non-immersive VRE and CT in Patients With Tennis Elbow
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/759
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Tennis Elbow
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group I (Experimental)
  Interventions: Diagnostic Test: traditional physiotherapy
- Interventional group II (Active Comparator)
  Interventions: Combination Product: Non-immersive VR therapy

INTERVENTIONS:
Diagnostic Test: traditional physiotherapy — Participants in this arm will undergo traditional physiotherapy exercises for managing tennis elbow.
  Arms: Interventional group I
Combination Product: Non-immersive VR therapy — Participants undergo a VR-based rehabilitation program targeting tennis elbow symptoms. Sessions last 30 minutes, conducted 3 times per week for 6 weeks. Exercises focus on improving grip strength, wrist flexibility, and functional movement through interactive VR environments that visually engage the affected arm, promoting adherence and motivation without full immersion. The VR setup includes headsets or screens that enable visual interaction, enhancing the rehabilitation experience. The goal is to alleviate pain, increase range of motion, and restore muscle strength.
  Arms: Interventional group II

SUMMARY:
This study investigates the comparative effectiveness of non-immersive virtual reality (VR) therapy and conventional physiotherapy in managing tennis elbow (lateral epicondylitis). Tennis elbow is a painful condition often characterized by chronic pain, reduced grip strength, and limited functionality.

DETAILED DESCRIPTION:
Conventional treatment approaches, including manual therapy and strengthening exercises, have been widely used but may not fully address the long-term rehabilitation needs of every patient. Virtual reality, an emerging tool in rehabilitation, has the potential to enhance patient engagement and adherence by providing an interactive therapeutic environment. Participants will be divided into two groups: one receiving VR therapy and the other conventional therapy, with each intervention lasting six weeks. Outcome measures include pain intensity (VAS), functional disability (DASH), patient satisfaction (PRTEE), grip strength, range of motion (ROM), and adherence rates. This study aims to determine if VR therapy can offer superior benefits over conventional

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25 to 50 years.
* Patient diagnosis with lateral epicondylitis.
* Patients that a medical doctor will be formally diagnosed to have tennis elbow, that is, lateral epicondylitis.
* Patients who have specific pain and function impairment associated with tennis elbow.
* Patients giving written consent to participate in the study. Willing to participate and provide informed consent.

Exclusion Criteria:

* Patients with neurological conditions whereby they have abnormal functioning of their arms.
* Any previous surgical intervention for tennis elbow The presence of other significant musculoskeletal diseases in the upper extremity Severe cardiovascular or neurological disorders.

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 12 Months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain.
Handheld Dynamometer | 12 Months
  This instrument is scored using force production in kilograms (0-90) or pounds (0-200). Standardized procedure for positioning of instrumen

CONTACTS AND LOCATIONS:
Locations (1):
- Samahni, Near thq hospital samahni azad kashmir, Kashmir, Azad Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No